CLINICAL TRIAL: NCT06130592
Title: Technical Feasibility Study of Ultrasound Muscle Imaging in Antenatal Ultrasound Screening of Congenital Multiple Arthrogryposis
Brief Title: Technical Feasibility Study of Ultrasound Muscle Imaging in Antenatal Ultrasound
Acronym: FetUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC21.0423
Record Dates: First submitted 2023-04-24; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Arthrogryposis Multiplex Congenita (AMC)
MeSH Terms: conditions — Arthrogryposis

STUDY DESIGN:
Intervention Model Description: study prospective,randomized ,two groups (low risk of AMC vs hight risk of AMC), multicentre
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high risk of Arthrogryposis AMC (Active Comparator): Patient with a diagnosis during the 1st, 2nd, or 3rd trimester ultrasound, of an abnormality of position / deformation of one or more joints, and / or an abnormality of fetal movements at screening ultrasound or interrogation
  Interventions: Diagnostic Test: ultrasound muscle imaging technique
- low risk of Arthrogryposis AMC (Active Comparator): Patient coming for screening ultrasound
  Interventions: Diagnostic Test: ultrasound muscle imaging technique

INTERVENTIONS:
Diagnostic Test: ultrasound muscle imaging technique — ultrasound muscle imaging technique in antenatal ultrasound screening of congenital multiple arthrogryposis

SUMMARY:
The objective of the study is to evaluate the performance of muscle ultrasound sections on antenatal ultrasound between 21-24 amenorrhea weeks for the screening of muscle atrophy, in a sample of low-risk and high-risk pregnancies of congenital multiple arthrogryposis

DETAILED DESCRIPTION:
Frequent rare diseases (100-200 births in France / year), congenital multiple arthrogryposis include a set of pathologies characterized by the limitation of joint movements at least two joint levels.Their functional prognosis and muscle atrophy are often severe after birth.

Routine ultrasound call signs are either non-specific or insensitive and difficult to detect due to time constraints. Antenatal ultrasound screening is not very effective for these pathologies, which are often particularly serious.

The main criterion will be the success rate of realization of all four ultrasound sections at the extremities (deltoide, biceps, quadriceps, triceps) and measurements of the distances "skin - muscle fascia" and "muscular fascia - periosteum" between 21-24 amenorrhea weeks

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman consulting in one of the two obstetric gynecology departments in connection with the CPDPN (Multidisciplinary Prenatal Diagnostic Centers) of the University hospitals of Lyon or Grenoble.
* Mono-embryonic pregnancy.
* Gestational ages retained on the first dating ultrasound or the 1st trimester ultrasound between 21-24 amenorrhea weeks.
* For women at "high risk": diagnosis during ultrasound of the 1st, 2nd, or 3rd trimesters, of an abnormality of position / deformation of one or more joints, and / or an abnormality of fetal movements on screening ultrasound or interrogation (population group at "high risk of AMC").
* Regulatory criteria: adults, affiliated to a social security scheme, having signed a consent

Exclusion Criteria:

* Multiple pregnancies, and / or non-progressive .
* Obese women (BMI > 30 in early pregnancy)
* Subject in a period of exclusion from another study
* Subject under administrative or judicial supervision
* Subject who cannot be contacted in case of emergency

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant woman
Enrollment: 230 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of achievement (success) of all four sections at the extremities | 72 hours +/- 24 hours
  Rate of achievement (success) of all four sections at the extremities for measurements (in mm) of the distances "skin - muscular aponeurosis" and "muscular aponeurosis- periosteum" between 21-24 amenorrhea weeks

SECONDARY OUTCOMES:
Rate of achievement (success) of each four sections | 72 hours +/- 24 hours
  Rate of achievement (success) of measurements (in mm) of the distances "skin - muscular aponeurosis" and "muscular aponeurosis- periosteum" between 21-24 amenorrhea weeks for biceps, deltoide, quadriceps and sural triceps
Collect the raisons for the failure of achievement of all sections | 72 hours +/- 24 hours
  Collect the raisons for the failure of achievement of all sections (Inadequate foetal position,Insufficient echogenicity, Reasons related to the position of the limbs (full extension or flexion of the elbows or knees, abduction of the shoulder, other), other raison (to be specified)
Duration of realization of the ultrasound sections | 72 hours +/- 24 hours
  Duration of realization of the ultrasound sections (investigators make an hypotheses of a duration of 3 minutes necessary for the realization of the sections
Comparison of the completion rates of all cuts during ultrasounds between high- and low-risk patients | 72 hours +/- 24 hours
  Comparison of the completion rates of all cuts during ultrasounds between high- and low-risk patients
Concordance of measures (CCI coefficient) will be evaluated in intra-observer and inter-observer respectively | 72 hours +/- 24 hours
  Concordance of measures (CCI coefficient) will be evaluated in intra-observer and inter-observer respectively by dividing by half the high-risk pregnancies, to whom it will be proposed a 2nd ultrasound of the 2nd trimester, within 3 days (±24) hours by the same / another referent sonographer in the same center. A group of 30 low-risk pregnancies will be evaluated in the same way, with the study of intra-observer reproducibility in 15. The sample of 30 pregnancies in which two measurements are made makes it possible to obtain a lower bound of the 95% confidence interval of the intra-class correlation coefficient greater than 0.7, if this coefficient is 0.85 or more. This threshold is usually considered to reflect a satisfactory concordance.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus DIETERICH, MD,PhD, Principal Investigator — Univ. Grenoble Alpes Inserm U1209 IAB CHU Grenoble Alpes